CLINICAL TRIAL: NCT04110574
Title: Computed Tomography Evaluation of Urinary Stones Densities Compared to in Vitro Analysis of Its Chemical Composition
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Somia Usama Mohamed Rabea, Resident doctor, Assiut University
Other Study IDs: CT of urinary stones densities
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Urinary Calculi
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ability to predict stone composition, which influences patient treatment, depends on the accurate measurement of CT attenuation of stones. We will study the effects of stone composition, stone size, and scan collimation width on the measurement of attenuation in vitro.

DETAILED DESCRIPTION:
Recently, the use of noncontrast spiral computerized tomography (NCCT) has gained widespread acceptance in the evaluation of urinary stone patients. It has long been used clinically to evaluate the causes of radiolucent filling defects using Hounsfield units (HU) to distinguish calculi from tumor or blood clots, and to identify nonurologic causes of flank pain (Smith R etal ). Urinary stones have a significantly higher CT attenuation than the surrounding soft tissues and are virtually always visible on NCCT. Knowing the composition of a urinary calculus is frequently a key factor in determining its most appropriate management. Should the urine be alkalinized? Will the stone be amenable to extracorporeal shock wave lithotripsy (ESWL), or should ureteroscopy or percutaneous lithotripsy be attempted? Different techniques have been used to assist in determining the correct chemical composition of calculi. Urine pH, urinary crystals, prior stone history and the presence of urea-splitting organisms (Ramakumar S,etal). Several in vitro studies have suggested that NCCT can demonstrate measured differences in radiodensity among different urinary stones (Mitchenson HD etal,).With these clinical problems in mind, we sought to determine whether the composition of urinary calculi could be predicted by their CT characteristics in an attempt to find out the best technique for distinguishing the various stones compositions, provided that it is clinically practical and would not require repeated imaging of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Any Age will be included .
* Patient with suspected or known urinary stone disease.
* Eligible for doing NCCT.
* Giving written consent to participate

Exclusion Criteria:

* Patient with classical NCCT contraindication like morbid obesity and pregnancy .
* Patients with urinary stones will be treated by ESWL
* Refusal participation .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected or known urinary stone disease and were included in the study who attend to out patient clinic of Urology department of Assiut university hospital or admitted in the ward.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
comparison of CT densities of urinary stones with its chemical composition | Baseline
  determination whether the composition of urinary calculi could be predicted by their CT characteristics in an attempt to find out the best technique for distinguishing the various stones compositions .

REFERENCES:
- See also: Determination of the chemical composition of urinary calculi by non contrast spiral computerized tomography. — https://www.ncbi.nlm.nih.gov/pubmed/?term=10.1007%2Fs00240-004-0454-2